CLINICAL TRIAL: NCT06271083
Title: A Parallel-group, Randomized Controlled Trial of Internet-based Behavior Therapy for Adults With Tourette Syndrome
Brief Title: Internet-based Behavior Therapy for Adults With Tourette Syndrome
Acronym: TICNET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ekaterina Ivanova, Postdoctoral researcher, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-06541-01
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Tourette Syndrome; Chronic Tic Disorder
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavior therapy with exposure and response prevention (Experimental)
  Interventions: Behavioral: Exposure with response prevention
- Psychoeducation with general psychological support (Active Comparator)
  Interventions: Behavioral: Brief psychoeducation with general psychological support

INTERVENTIONS:
Behavioral: Exposure with response prevention — The central component of the intervention will be ERP. During the treatment, participants will receive information about tics and how to work with ERP. Continuously throughout the treatment patients will work with exposing themselves to situations that trigger their premonitory urges and practice suppressing their tics. They will learn different strategies to provoke their premonitory urges to make suppression of their tics more challenging and gradually increase the time they can suppress the tics. A central tool in the treatment will be the Ticstimer, a worksheet where patients will continuously record their ERP practice, and the time they manage to suppress tics. The patients will be encouraged to work with the Ticstimer daily.
  Arms: Behavior therapy with exposure and response prevention
Behavioral: Brief psychoeducation with general psychological support — Participants who are randomized to the control group will receive access to brief psychoeducational content in the platform in combination with general psychological support from a therapist. No active BT components (BT, Habit Reversal Training, applied relaxation) are provided to the participants in the control group. The therapists will welcome the patients to the treatment, encourage them to engage in the treatment content and reach out to the therapist if they have any questions. Thereafter, the therapists will only reply to the patients' messages without taking any contact initiative themselves (unless there is an indication of severe deterioration or severe depressive symptoms or suicidal ideation requiring medical attention)
  Arms: Psychoeducation with general psychological support

SUMMARY:
This study protocol outlines a parallel-group, randomized controlled trial (RCT) designed to evaluate the effectiveness of Internet-delivered behavior therapy (BT) based on exposure with response prevention (ERP) for adults with Tourette syndrome (TS) or chronic tic disorder (CTD). The primary aim is to evaluate the effects of Internet-delivered ERP-based BT on tic severity compared to a control condition offering general psychological support at week 11 counting from the treatment start. The primary outcome measure is the Yale Global Tic Severity Scale - Total Tic Severity subscale (YGTSS-TTS). Secondary outcomes include measures of tics-related impairment, work and social adjustment, rates of responders, self-rated tic severity, symptoms of depression, and quality of life. Long-term maintenance of results will be assessed at week 23 and 14 months after the treatment start. Participants will be recruited nationwide. The intervention group will receive 10 weeks of ERP-based therapy delivered through an online platform, with therapist support. The control group will receive psychoeducational content and general psychological support. Adherence to treatment, adverse events, and patient safety will be closely monitored throughout the trial. The study population will be intent-to-treat and the between-group differences at the primary endpoint will be assessed using an analysis of covariance (ANCOVA) with pre-score of the measure as covariate. A health-economic evaluation will assess the cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years of age.

Primary diagnosis of TS/CTD, according to criteria in Diagnostic and Statistical Manual of mental disorders 5th edition.

Provided digital informed consent.

Have a Total Tic Severity Score (TTS) of >15, or >10 for individuals with motor or vocal tics only, in the past week, as measured by the Yale Global Tic Severity Scale (YGTSS).

Being willing and able to follow the study procedures and participate in the 10-week treatment program.

Being fluent in Swedish.

Have regular access to a computer connected to the Internet, sufficient technical skills to use the treatment platform, as well as a mobile phone to receive text messages.

Exclusion Criteria:

Ongoing or planned psychological treatment for TS/CTD.

Previous BT for tics of a minimum of 8 sessions with a qualified therapist within 12 months prior to assessment.

Adjustment of medication for tics within the last two months prior to assessment.

Severe psychiatric comorbidities such as organic brain disorders, bipolar disorder, ongoing psychosis, anorexia nervosa or substance use disorders that can interfere with the treatment for TS/CTD.

Acute psychiatric problems such as severe depression or suicidal risk needing immediate psychiatric care.

Severe tics causing immediate risk to the participants themselves or to others and requiring urgent medical attention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale - Total Tic Severity subscale (YGTSS-TTS) | Baseline, week 11 (primary end-point), 23 and 14 months after the treatment start.
  The YGTSS is made up of a semi-structured interview, followed by a questionnaire where individuals are asked to rate the severity of their tic symptoms (both motor and vocal) in domains such as: number, frequency, intensity, complexity, and interference. The Total Tic Severity subscale has a range of 0-50. A higher score suggests higher tic severity.

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) - impairment scale | Baseline, week 11 (primary end-point), 23 and 14 months after the treatment start.
  The YGTSS is made up of a semi-structured interview, followed by a questionnaire where individuals are asked to rate the severity of their tic symptoms (both motor and vocal) in domains such as: number, frequency, intensity, complexity, and interference. There is also an impairment scale, where the individual rates how the tic impacts on their daily life and activities. The impairment score has a range of 0-50 (steps of 0,10,20,30,40,50). A higher score suggests or a greater impact the tics have on the person's life.
Clinical Global Impression (CGI) | Baseline, week 11 (primary end-point), 23 and 14 months after the treatment start.
  The Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) Scales will be used to assess overall clinical severity and consequent treatment response (scores of "very much improved" (1) or "much improved" (2) will define treatment response according to previous trials in tic disorders.
Gilles de la Tourette Syndrome Quality of Life Scale (QTS-QoL) | Baseline, week 11 (primary end-point), 23 and 14 months after the treatment start.
  QTS-QoL is a syndrome-specific quality of life scale with 27 items scored on a 5-point likert scale from no problems to very severe problems.The total score ranges from 0 to 108 with higher score indicating more severe problems.
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, week 3, 7, 11 (primary end-point), 23 and 14 months after the treatment start.
  MADRS is a 9-item depressive symptoms scale where the symptoms are assessed on a 7-point likert scale from no symptoms to very high severity. The total score ranges from 0 to 54 with higher score indicating more severe problems.
Adult Tic Questionnaire (ATQ) | Baseline, week 2-10, week 11 (primary end-point), week 23 and 14 months after the treatment start.
  The Adult Tic Questionnaire (ATQ) is a self-report measure used to assess the frequency, severity, and impact of tic symptoms in adults with Tourette syndrome or chronic tic disorder. It includes questions on 28 different types of tics, each type being scored regarding both intensity and frequency using 4-step likert-scale. The total score ranges between 0 and 224 with higher scores indicating higher tic severity.
Work and social adjustment scale (WSAS) | Baseline, week 2-10, week 11 (primary end-point), week 23 and 14 months after the treatment start.
  Work and social adjustment scale (WSAS) includes five questions on the person's functioning at home, school/work, leisure, relationships and social activities, each scored on a 9-step likert scale. The total score ranges between 0 and 40 with higher scores indicating lower functioning.
Treatment Inventory of Costs in Psychiatric Patients (TIC-P) | Baseline, week 11 (primary end-point), 23 and 14 months after the treatment start.
  Self-rated questionnaire on healthcare utilization and productivity losses in patients with a psychiatric disorder. The TIC-P questionnaire measures costs in two dimensions: use of health resources and loss of productivity. Lower cost is better.
Assessing Quality of Life 6 Dimensions (AQoL-6D) | Baseline, week 11 (primary end-point), 23 and 14 months after the treatment start.
  Used to assess cost-effectiveness. 20 questions that assess different aspects of quality of life. The AQoL provides a utility score that ranges from 1.00 (full health) to 0.00 (death-equivalent health states) to -0.04 (health states worse than death).

OTHER OUTCOMES:
Internet Intervention Patient Adherence Scale for Guided Internet-Delivered Behavioural Interventions (iiPAS) | At week 6 and 11 after the treatment start
  The iiPAS is a 5-item, clinician-rated measure of patient adherence to internet-delivered behavioral interventions. The 5 items are rated by treating clinicians and cover 5 central aspects of adherence: the patient's work pace, engagement, communication with the clinician, motivation for change, and login frequency. The clinicians assess each domain on a 5-point likert scale (scored 0-4), with a total score ranging between 0-20 where higher score indicates higher treatment adherence.
Credibility/Expectancy Questionnaire (CEQ) | At treatment week 5
  Measures treatment expectancy and rationale credibility. The CEQ is a 5-item measure of the treatment's credibility and the patients' expectations. The patients assess each domain on a 11-point likert scale (scored 0-10), with a total score ranging between 0-50 where higher score indicates higher credibility and higher expectations.
Working Alliance Inventory-Short Form Revised (WAI-SR) | At treatment week 5
  Measures the therapeutic alliance in therapy. The WAI-SR is a 12-item measure of the patient's experience of their working alliance with the therapist. The patients assess each item on a 7-point likert scale (scored 0-6), with a total score ranging between 0-72 where higher score indicates higher better working alliance according to the patient.
Checklist for negative events | At week 11 (primary end-point) and 23.
  A checklist listing 16 different negative events asking about how often the participant experienced each of them and whether the participant thinks the event was due to the treatment they received.
Events during treatment and adverse events | At week 3, 7, 11 (primary end-point) and 23.
  Three questions on whether the participant needed to seek more care, change their medication, start another treatment or be treated in inpatient care.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Ivanova, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Sannemalm M, Lybert N, Gunnarsson L, Andren P, Kraepelien M, Bragesjo M, Fondberg R, Ivanov VZ, Mataix-Cols D, Fernandez de la Cruz L, Andersson E, Ruck C, Ivanova E. Study protocol for a parallel-group randomized controlled trial of internet-delivered behavior therapy for adults with Tourette syndrome. Front Digit Health. 2025 Aug 29;7:1518666. doi: 10.3389/fdgth.2025.1518666. eCollection 2025. PMID 40949315